CLINICAL TRIAL: NCT05181358
Title: Evaluation of the Relationship Between Different Postoperative Analgesia Techniques and Post-cesarean Quality of Recovery; Prospective Observational Study
Brief Title: Relationship Between Analgesia Techniques and Post-cesarean Recovery Quality
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Other Study IDs: ObsQoR-10 PNB
Record Dates: First submitted 2021-12-19; First posted 2022-01-06 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Quality of Recovery; Cesarean Section
Keywords: Quality of recovery; ObsQoR-10; regional analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The question remains whether the patients in whom USG-guided regional anesthesia and analgesia techniques are applied have a better recovery score than subarachnoid morphine administration, which is considered the gold standard. The primary aim of this study is to evaluate the quality of recovery score using the Obstetric Recovery Quality Score-ObsQoR-10 questionnaire experienced by the patients who underwent elective cesarean section and compare the results of different regional anesthesia techniques with subarachnoid morphine.

DETAILED DESCRIPTION:
National and international guidelines, hospital protocols, the anesthesiologist's experience, and the patient's decision play a role in selecting the technique used for postoperative analgesia after cesarean section. The quality of recovery score experienced following elective cesarean section in a total of 180 patients over one year (December 31, 2021-2022) who applied subarachnoid morphine, lateral TAP block, posterior-TAP block, QL block, ESP block, and TFD block (30 patients for each technique) will be evaluated with the ObsQoR-10 questionnaire 24 hours after delivery. The regional anesthesia techniques information applied to the patients will be obtained from the patient file. Researchers will not perform any interventional procedure, and any randomization will not be applied. After the data collection process for the study is completed, ObsQoR-10 will be compared statistically. The secondary aims of this study are to compare the cases in terms of postoperative analgesia and antiemetic requirements, first food intake and standing up without support, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Term obstetric patients aged 18-47 years who underwent elective cesarean section under spinal anesthesia and applied regional anesthesia techniques such as lateral TAP, posterior-TAP, QL, ESP, and TFD blocks or subarachnoid morphine.

Exclusion Criteria:

* Patients with psychiatric disorders
* Patients requiring emergency cesarean section.
* Patients with additional obstetric pathology (such as placenta previa, preeclampsia, DM)
* The need for intensive care in the mother or newborn at the end of the birth.
* Patients who have undergone general anesthesia.
* Preterm pregnants

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only the patients who underwent elective cesarean section will be recruited
Study Population: Term obstetric patients who underwent elective cesarean section under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Obstetric Quality of Recovery | The first 24 hours postoperatively
  Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool

CONTACTS AND LOCATIONS:
Locations (1):
- Betul Kozanhan, Konya, Turkey (Türkiye)